CLINICAL TRIAL: NCT00789724
Title: Recombinant Human Interleukin-1 Receptor Antagonist, Anakinra, to Prevent Post-infarction Remodeling: the Virginia Commonwealth University Anakinra Remodeling Trial (VCU-ART)
Brief Title: Anakinra to Prevent Post-infarction Remodeling
Acronym: VCU-ART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VCU-ART
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Results first posted 2010-08-24 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: ST Segment Elevation Acute Myocardial Infarction
Keywords: acute myocardial infarction
MeSH Terms: interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anakinra (Experimental): Anakinra 100 mg given daily by subcutaneous injection for 14 days
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): 0.67 ml of NaCl 0.9% solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra — 100 mg daily subcutaneous injection for 14 days
  Other Names: Kineret (TM)
  Arms: Anakinra
Drug: Placebo — 0.67 ml of NaCl 0.9% subcutaneously daily for 14 days
  Arms: Placebo

SUMMARY:
Thousands of patients die daily from early and late complications of a heart attack (acute myocardial infarction, AMI). Patients surviving AMI remain at high risk of death from adverse cardiac remodeling (dysfunction and enlargement of the heart) leading to heart failure (weakening of the heart).

Current interventions proven to reduce adverse remodeling and progression to heart failure include early reperfusion (restoring blood flow to the heart muscle) and long-term use of medicines that block the effects of hormones (such as angiotensin II, norepinephrine and aldosterone) involved in adverse remodeling. Despite these treatments, however, many patients continue to develop heart failure within 1 year of AMI. These patients are at very high risk of death.

Numerous changes occur in the hearts of patients after AMI that lead to adverse remodeling. Ischemia (lack of oxygen) and infarction (cell damage) lead to increased interleukin-1 (IL-1) production in the heart. IL-1 plays a critical role in adverse cardiac remodeling by coordinating the inflammatory pathway (leading to wound healing) and apoptotic pathway (leading to cell death).

In opposition to IL-1 activity, the human body produces a natural IL-1 receptor antagonist that blocks the effects of IL-1. The drug form of this IL-1 receptor antagonist (anakinra) is currently FDA approved for the treatment of rheumatoid arthritis, an inflammatory disease characterized by excessive IL-1 activity. Experimental studies show that anakinra is able to prevent cardiac remodeling and improve survival in mice after AMI.

We hypothesize that anakinra will show similar benefits in human patients by preventing adverse remodeling and heart failure after AMI.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Acute (<24 hours) onset of chest pain
* New or presumably new ST elevation on ECG
* Planned coronary angiography for percutaneous revascularization

Exclusion Criteria:

* Inability to give informed consent
* Late presentation (>24 hours)
* Unsuccessful revascularization or urgent coronary bypass surgery
* Hemodynamic instability
* End-stage congestive heart failure (AHA/ACC stage C/D, NYHA class IV)
* Preexisting severe LV dysfunction (LVEF<20%) or severe valvular disease
* Severe asthma
* Pregnancy ( pre-enrollment pregnancy test)
* Contraindications to cardiac MRI or cardiac angiography
* Severe coagulopathy (INR>2.0, Platelet count<50,000/mm3)
* Severe renal insufficiency (creatinine clearance <30 ml/min/m2)
* Recent (<14 days) use of anti-inflammatory drugs (NSAIDS excluded)
* Chronic inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Denicolai M, Morello M, Golino M, Corna G, Del Buono MG, Agatiello CR, Van Tassell BW, Abbate A. Interleukin-1 Blockade in Patients With ST-Segment Elevation Myocardial Infarction Across the Spectrum of Coronary Artery Disease Complexity. J Cardiovasc Pharmacol. 2025 Mar 1;85(3):200-210. doi: 10.1097/FJC.0000000000001652. PMID 39531530
- [Derived] Del Buono MG, Damonte JI, Chiabrando JG, Markley R, Turlington J, Trankle CR, Kang L, Biondi-Zoccai G, Van Tassell BW, Abbate A. Effect of IL-1 Blockade With Anakinra on Heart Failure Outcomes in Patients With Anterior Versus Nonanterior ST Elevation Myocardial Infarction. J Cardiovasc Pharmacol. 2022 Jun 1;79(6):774-780. doi: 10.1097/FJC.0000000000001240. PMID 35170493
- [Derived] Abbate A, Kontos MC, Abouzaki NA, Melchior RD, Thomas C, Van Tassell BW, Oddi C, Carbone S, Trankle CR, Roberts CS, Mueller GH, Gambill ML, Christopher S, Markley R, Vetrovec GW, Dinarello CA, Biondi-Zoccai G. Comparative safety of interleukin-1 blockade with anakinra in patients with ST-segment elevation acute myocardial infarction (from the VCU-ART and VCU-ART2 pilot studies). Am J Cardiol. 2015 Feb 1;115(3):288-92. doi: 10.1016/j.amjcard.2014.11.003. Epub 2014 Nov 13. PMID 25482680

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started in November 2008. During the first 4 months, 33 patients admitted with STEMI were screened and 10 patients were enrolled. One patient withdrew consent to the study on day 2 prior to all assessment and was excluded. The Institutional Review Board then approved enrollment of an additional patient who was enrolled in May 2009.
Period: Overall Study
Arm/Group | Anakinra | Placebo
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anakinra | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (13) | 52 (15) | 48 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Difference Between the Anakinra Arm and Placebo Arm in Change in End-systolic Volume Indices From Baseline to Follow up Exam 10-14 Weeks Later at Cardiac Magnetic Resonance Imaging.
Time Frame: 10-14 weeks
Measure: Median (Inter-Quartile Range); unit: mL/m2
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 5 | 5
mL/m2 | -3.2 [-4.5 to -1.2] | 2.0 [1.0 to 11.0]
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority or Other; p = 0.033, ANOVA

2. Other Pre Specified Outcome: Difference Between the 2 Arms in the Percentage of Patients With Any of the Following : a) End-systolic or End-diastolic Volume Index Increase >10%; b) Ejection Fraction Decrease >10%; c) E/E'>15 at Follow up
Time Frame: 10-14 weeks
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Difference Between the 2 Arms in Change in the Number of Circulating Endothelial Progenitor Cells From Baseline to Follow up Exam
Time Frame: 10-14 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Difference Between the 2 Arms in Change in Serum BNP Levels, C-reactive Protein, and Hemoglobin A1c% From Baseline to Follow up
Time Frame: 10-14 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Difference Between the 2 Arms in the Incidence of Significant Cardiac Arrhythmias in the Acute Phase
Time Frame: 48 hours
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Difference Between the 2 Arms in the Number of Adverse Effects Including a) All Events; b) All Events Requiring Unblinding of the Treatment; c) All Events Requiring Early Termination of the Intervention
Time Frame: 10-14 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Difference Between the 2 Arms in Change in Oxygen Uptake Kinetics From Baseline to Follow up Exam at Submaximal Cardiopulmonary Exercise Test
Time Frame: 10-14 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Difference Between the 2 Arms in Change in E/E' Ratios and Myocardial Performance (Tei) Indices From Baseline to Follow up Exam at Transthoracic Echo-color-Doppler Cardiac Exam
Time Frame: 10-14 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Difference Between the 2 Arms in Change in End-diastolic Volume Indices and Ejection Fraction Values From Baseline to Follow up Exam at Cardiac Magnetic Resonance Imaging
Time Frame: 10-14 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Anakinra | Placebo
Serious Adverse Events (participants affected / at risk) | 2/5 | 4/5
Other Adverse Events (participants affected / at risk) | 2/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (N=5) | Placebo (N=5)
Recurrent acute coronary syndrome (Cardiac disorders) | 2 (2) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (N=5) | Placebo (N=5)
Injection site pain (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No